CLINICAL TRIAL: NCT06526832
Title: A Phase 1, Dose-Escalation and Dose-Expansion Study Evaluating the Safety, Tolerability and Efficacy of BST02 in Treating Locally Advanced Liver Cancer
Brief Title: A Phase 1 Study of BST02 in Treating Locally Advanced Liver Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioSyngen Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSG-BST02-01
Record Dates: First submitted 2023-09-06; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Liver Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BST02 (Experimental): Patients who receive BST02 infusion.
  Interventions: Biological: BST02

INTERVENTIONS:
Biological: BST02 — BST02 is a tumor infiltrating lymphocyte product manufactured from the sample collected in the patient's tumor lesion.

SUMMARY:
The goal of this clinical trial is to investigate the BST02, a tumor infiltrating lymphocyte product, collected from the locally advanced liver cancer subjects

The main questions it aims to answer are:

1. Safety and tolerability of BST02.
2. Preliminary efficacy of BST02. Participants will receive a cytoreductive surgery to collect samples for the manufacture of BST02.

Participants will receive BST02 infusion followed by IL-2 infusion. Blood samples will be collected for the analysis of PK and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years (inclusive);
2. Patients with histologically or cytologically confirmed advanced liver cancer (including hepatocellular carcinoma and intrahepatic cholangiocarcinoma) staged according to the Barcelona Clinic Liver Cancer (BCLC) Classification Criteria as stage C or stage B unsuitable for local treatment/progression on local treatment; or intrahepatic cholangiocarcinoma that is unresectable, recurrent, or metastatic (AJCC 2017, 8th edition, TNM staging of stage IV).
3. Failure (disease progression or intolerability) after at least first-line guideline-recommended systemic therapy (Atezolizumab + Bevacizumab, Sintilimab + Bevacizumab analogs; Donafenib, Lenvatinib, Sorafenib; FOLFOX4; Gemcitabine in combination with Cis-platin, etc.), refused to receive the standard systemic therapy by the subject, or deemed inappropriate for standard systemic therapy by the investigator;
4. At least one surgically resectable tumor lesion that has not received radiation therapy or other local treatment within 28 days which will be used to prepare BST02 cells;
5. At least one measurable lesion in line with the definition of mRECIST criteria after TIL sampling surgery. If the target lesion is intrahepatic, arterial phase enhancement imaging is required;
6. Eastern Cooperative Oncology Group (ECOG) score≤1;
7. Child-Pugh score for hepatic cirrhosis ≤7;
8. Expected survival time≥3 months;
9. Adequate organ and bone marrow functions, as defined below, at the time of assessment during the screening and preparation period (within 14 days prior to TIL sampling):

   Hematology: Absolute Neutrophil Count (ANC)≥1.5×109/L, Blood Platelet Count (PLT)≥90×109/L, Hemoglobin (HGB)≥80 g/L (no transfusion or erythropoietin treatment within 14 days); Hepatic function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) levels≤5 × Upper Limit of Normal (ULN); Serum Total Bilirubin (TBil) ≤ 1.5×ULN; if Gilbert's syndrome is diagnosed: TBil ≤ 3×ULN; Coagulation function: Activated partial thromboplastin time (APTT) ≤ 1.5×ULN, while International Normalized Ratio (INR), Prothrombin Time (PT) ≤ 1.5×ULN; Renal function: Serum creatinine (Cr)≤1.5×ULN or Creatinine Clearance (Ccr) ≥ 60mL/min (Cockcroft-Gault formula); Cardiac function test: Left Ventricular Ejection Fractions (LVEF)≥50% by echocardiography; arrhythmia with no need for treatment, Fridericia QT correction formulas (QTcF)≤470 ms (QTcF is calculated using the Fridericia formula, i.e., QTcF = QT/(RR^0.33), RR is the standardized heart rate value, RR=60/heart rate; if the results of the first test are abnormal, the test can be repeated twice at an interval of at least 5 minutes and the comprehensive result/mean value should be considered to determine the eligibility); Lung function: Percentage of FEV1 to the predicted value (FEV1%) ≥ 60%;
10. Prior treatment-induced adverse reactions have recovered to ≤ grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) 5.0 (except for toxicities such as alopecia, grade 2 or less peripheral neurotoxicity, and other toxicities that do not pose a safety risk as determined by the investigator) prior to TIL sampling;
11. Subjects agree to use effective contraceptives from the time of signing the informed consent form until 6 months after infusion of BST02 cells (non-drug measures for contraception must be taken);
12. Subjects should fully understand the trial and voluntarily sign the informed consent form, and be able to comply with the visits and related procedures specified in the protocol.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects with a prior history of severe allergy and hypersensitivity to the investigational drugs including, but not limited to, cyclophosphamide, fludarabine, IL-2, and the components of BST02;
3. Subjects with prior or current history of hepatic encephalopathy; patients with known central nervous system metastases uncontrolled by other treatment or untreated; with exception of patients who have stabilized their symptoms after treatment, and discontinued the treatment of glucocorticoid and anticonvulsant medications ≥4 weeks prior to lymphodepletion preconditioning;
4. Presence of clinically significant ascites, defined as: Positive signs of ascites on physical examination or ascites that needs to be controlled with interventional therapy (only those with ascites on imaging without intervention may be included); (5) The Indocyanine Green retention test after 15 min (ICG-R15) is ≥30%;

(6) History of organ transplantation, hematopoietic stem cell transplantation; (7) Other serious medical conditions that may limit the subject's participation in this trial, including but not limited to: Hypertension that is uncontrolled by medication (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at rest after taking medication); Uncontrolled diabetes: Fasting blood glucose levels remain above 1 mmol/L after standardized treatment with insulin; Unstable cardiovascular diseases: Uncontrolled congestive cardiac failure, infarct myocardial or unstable arrhythmia or unstable arrhythmia within the last 6 months, percutaneous coronary interventional procedure, acute coronary syndromes, coronary artery bypass transplant; cerebrovascular accident, transient ischemic attack, cerebral embolism, deep vein thrombosis, etc.; Uncontrolled respiratory system disorder: Pulmonary embolism, chronic obstructive pulmonary disease, interstitial lung disease, etc.; Active, autoimmune diseases requiring systemic therapy during the period of the study: Subjects with eczema, vitiligo, psoriasis, alopecia, or Graves's disease who do not require systemic treatment within the last 2 years, other autoimmune disorders that are not expected to recur, and subjects with type I diabetes mellitus who require only insulin replacement therapy may be enrolled; Active infection or active tuberculosis infection with a need for systemic therapy; Mental illness, except for mild depression, and other mild conditions; (8) Patients who are HIV-positive, or positive for syphilis spirochete antibodies; Patients with active hepatitis B or C are required to adopt antiviral therapy during the whole study. Active hepatitis B is defined as positive hepatitis B core antibody (HBcAb) or hepatitis B surface antigen (HBsAg) and HBV-DNA >2000 IU/ml. Active hepatitis C is defined as HCV RNA above the lower limit of detection; (9) Subjects have taken any immunosuppressive drugs, such as corticosteroids, within 4 weeks prior to TIL sampling or had combined diseases needing application of immunosuppressive medications for the duration of the trial as judged by the investigator. However, physiologic doses of glucocorticoids (i.e., a maximum dose of 15 mg/day for prednisone or an equivalent dose of other glucocorticoids) are permitted, and inhalational, intranasal, topical, or prophylaxis use of corticosteroids are allowed against contrast allergy; (10) Subjects who have received anti-PD-1/ PD-L1 monoclonal antibody treatment within 4 weeks prior to lymphodepletion preconditioning , or undergone local treatments such as surgery (except BST02 sampling surgery), interventional therapy, radiotherapy, ablation, or systemic therapy against liver cancer (including those who participated in other clinical trials of drug therapy; metabolism of drugs with 5 half-lives of less than 4 weeks, whichever is shorter); or immunotherapy such as thymopeptide, interferon, or any traditional Chinese medicine used for tumor control within 1 week prior to lymphodepletion preconditioning ; (11) Subjects who have received a live vaccine within 3 months prior to screening or planned to receive a live vaccine during the trial; (12) Subjects who have undergone major surgery within 4 weeks prior to screening or planned to receive surgery during the trial period (except for TIL sampling surgery); (13) Patients with surgical complications or delayed wound healing prior to lymphodepletion preconditioning who, in the judgment of the investigator, will be at increased risk for lymphodepletion, TIL therapy, IL-2 adjuvant therapy, or infection; (14) Subjects who have diagnosed as combined other primary malignant neoplasm within 5 years prior to screening, excluding radically treated basal cell carcinoma of skin, squamous cell carcinoma of skin, and/or radically resected carcinoma in situ; (15) Subjects who have received cell therapy products 6 months prior to lymphodepletion preconditioning; (16) Subjects with known alcoholism, drug or substance abuse, and others who, in the opinion of the investigator, are not suitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Occurence and incidence of adverse event and severe adverse events. | From the infusion (D0) to D28
  The occurrence and incidence (%) of Adverse Events (AEs) as well as Severe Adverse Events (SAEs) after infusion of BST02 for subjects in each dosing group
Maximum Tolerated Dose (MTD) and Dose-Limiting Toxicity (DLT) | From the infusion (D0) to D28
  The highest dose which the patients can tolerate, and the occurence of DLT events.

SECONDARY OUTCOMES:
Tumor response and survival. | From the infusion (D0) to D672 (2 years)
  Including following outcomes: Objective Response Rate (ORR), Disease Control Rate (DCR), Time to Response (TTR), Duration of Response (DOR), Progression-Free Survival (PFS), Overall Survival (OS). The tumor responses are judged according to mRECIST criteria.
PK parameter collection | From before infusion (D-2) to D28
  PK testing indicator for BST02: Peripheral blood CXCR3+CD8+ T-lymphocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Yaojun Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No